CLINICAL TRIAL: NCT05954078
Title: Circulating Tumor DNA Methylation Guided Postoperative Adjuvant Chemotherapy for High-risk Stage II/III Colorectal Cancer: A Multicenter, Prospective, Randomized Controlled Cohort Study (FINE Trial)
Brief Title: Circulating Tumor DNA Methylation Guided Postoperative Adjuvant Chemotherapy for High-risk Stage II/III Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Junjie Peng, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FINE Trial
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: High-risk Stage II Colorectal Cancer; Stage III Colorectal Cancer; Circulating Tumor DNA Methylation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mFOLFIRINOX adjuvant chemotherapy (Experimental): Patients will receive mFOLFIRINOX once every two weeks for 6 cycles as adjuvant chemotherapy, after which a blood test is conducted to check the status of ctDNA. If the ctDNA remains positive, the treatment continues for another 6 cycles. If the ctDNA becomes negative, then maintenance chemotherapy with single-agent capecitabine is given once every 21 days for 4 cycles.
  Interventions: Drug: mFOLFIRINOX adjuvant chemotherapy
- mFOLFOX6/XELOX adjuvant chemotherapy (Active Comparator): Patients will receive mFOLFOX6 once every two weeks for 6 cycles or XELOX once every three weeks for 4 cycles as adjuvant chemotherapy. After the treatment, a blood test is conducted to check the status of ctDNA. If the ctDNA remains positive, the treatment continues with another 6 cycles of mFOLFOX 6 or 4 cycles of XELOX given once every 21 days. If the ctDNA becomes negative, then maintenance chemotherapy with single-agent capecitabine is given once every 21 days for 4 cycles.
  Interventions: Drug: mFOLFOX6/XELOX adjuvant chemotherapy

INTERVENTIONS:
Drug: mFOLFIRINOX adjuvant chemotherapy — mFOLFIRINOX (oxaliplatin 85 mg/m2, irinotecan 180 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1) for 6 cycles
  Other Names: Oxaliplatin; Irinotecan; Leucovorin; 5-Fluorouracil
  Arms: mFOLFIRINOX adjuvant chemotherapy
Drug: mFOLFOX6/XELOX adjuvant chemotherapy — mFOLFOX6 (oxaliplatin 85 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 400mg/m2 infusion, and 2400mg/m2 as a 46-hour continuous infusion on day 1) for 12 cycles or XELOX (oxaliplatin 130mg/m2, ivgtt, Q3w; capecitabine 1000mg/m2, p.o, Q3w) for 8 cycles
  Other Names: Oxaliplatin; Leucovorin; 5-Fluorouracil
  Arms: mFOLFOX6/XELOX adjuvant chemotherapy

SUMMARY:
Colorectal cancer (CRC) is one of the most common gastrointestinal tumors. According to the latest cancer report, the incidence and mortality rates of CRC are both ranked top 5 among malignant tumors worldwide and continue to rise. Patients who receive treatment in the early stage (stage I) have a 5-year survival rate of approximately 90%. However, for high-risk stage II and III colorectal cancer patients, the 5-year survival rate is only 40%-70%, and almost half of the patients experience postoperative recurrence and metastasis.

Evidence suggests that Stage III CRC patients can benefit from standard adjuvant chemotherapy. It is worth noting that some high-risk stage II patients, especially those with T4N0, have a poorer prognosis compared to stage IIIA (T1-2N+). Adjuvant chemotherapy is now also recommended for postoperative cases of high-risk stage II CRC. Given the high effectiveness of the three-drug FOLFOXIRI regimen in treating metastatic CRC and the success of adjuvant chemotherapy in treating pancreatic cancer, the combination of 5-fluorouracil, oxaliplatin, and irinotecan may have a synergistic effect.

Extensive study results have shown that: (a) The status of ctDNA methylation after surgery is significantly correlated with patient prognosis, and patients who are positive for ctDNA methylation in the first 1-4 weeks after surgery (before adjuvant chemotherapy) have a poor prognosis. (b) Patients who are ctDNA methylation positive in the first 1-4 weeks after surgery (before adjuvant chemotherapy) can benefit from adjuvant chemotherapy, and achieving ctDNA methylation negativity through adjuvant chemotherapy significantly improves patient prognosis. This project focuses on exploring the optimized mode of postoperative adjuvant chemotherapy for high-risk stage II and III CRC guided by ctDNA methylation, which has high scientific and innovative value.

This multicenter, prospective, and randomized controlled cohort study uses a single-tube methylation-specific quantitative PCR (mqMSP) detection, which detects 10 different methylation markers and can quantitatively analyze plasma samples containing tumor DNA as low as 0.05%. This study will use this ctDNA methylation detection technology to perform quantitative detection of ctDNA methylation in the plasma of enrolled patients, and explore the effect of different chemotherapy regimens on ctDNA clearance rate and the prognostic value for ctDNA positive patients. We hope to screen out high-risk populations for recurrence through postoperative ctDNA testing, and administer more intensive chemotherapy regimens (chemotherapy upgrading) as early as possible to improve ctDNA clearance rate and patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

Patients who have been histopathologically diagnosed with colorectal adenocarcinoma;

Patients who have undergone radical curative resection of the primary tumors;

Patients with CRC of high-risk stage II and stage III based on final findings (UICC TNM Classification, 8th Edition);

Patients who tested positive for ctDNA methylation at 5-7 days after surgery prior to enrollment;

Patients with no obvious relapse confirmed by chest, abdominal, and pelvic CT scans, etc.;

Patients aged ≥ 18 and ≤80 years old, regardless of gender;

Patients with expected survival of more than 12 months;

Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1;

Patients who have no severe disorder in major organs (such as the bone marrow, heart, lungs, liver, and kidneys) and meet the following criteria: Neutrophil count ≥ 1,500/mm3, Platelet count ≥ 100,000/mm3, Hemoglobin ≥ 8.0 g/dL, Serum creatinine ≤ 1.5 mg/dL, Total bilirubin ≤ 1.5 mg/dL, ALT and AST ≤ 100 U/L

Patients with no diarrhea or stomatitis of Grade 2 or severer according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0;

Patients who voluntarily gave written consent to participate in the trial after receiving a thorough explanation of the trial before enrolling in the trial

Exclusion Criteria:

Neoadjuvant therapy performed before operation;

Blood transfusion performed during operation or within 2 weeks before operation;

Incomplete baseline samples, including preoperative plasma samples and plasma samples 5-7 days after operation;

Pregnant or lactating women who have fertility and do not take adequate contraceptive measures;

Have a history of other malignant tumors within 5 years, except cured cervical carcinoma in situ or non melanoma skin cancer;

Primary brain tumor or central nerve metastasis is not under control, with obvious intracranial hypertension or neuropsychiatric symptoms;

Patients with the following serious or uncontrollable diseases: severe heart disease, the condition is still unstable after treatment, including myocardial infarction, congestive heart failure, unstable angina pectoris, pericardial effusion with obvious symptoms or unstable arrhythmia within 6 months before enrollment; definite neuropathy or psychosis, including dementia or seizures; severe or uncontrolled infection; active disseminated intravascular coagulation and obvious bleeding tendency;

Significant impairment of important organ function;

Other conditions in which the investigator believes that the patient should not participate in this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
ctDNA clearance rate | ctDNA clearance rate after 3 months of chemotherapy (6 cycles or 4 cycles for chemotherapy); ctDNA clearance rate after 6 months of chemotherapy (12 cycles or 8 cycles for chemotherapy)
  The rate of ctDNA positive before chemotherapy that turns negative after adjuvant chemotherapy

SECONDARY OUTCOMES:
Disease-free survival (DFS) | Up to 3 years
  Defined as the time from randomization to relapse or death, whichever occurred first
Overall survival (OS) | Up to 5 years
  Overall Survival (OS) is defined as the time from the date of randomization to the date of documented death from any cause
Incidence of Adverse Events | Up to 3 years
  For each of the AEs due to the following study treatment, the frequency of cases with the worst grade in all courses according to CTCAE v5.0 will be calculated using all treated patients as the denominator.
Treatment Completion Rate | Up to 3 years
  This rate will be calculated for each eligible subject in accordance with the following equation. Treatment completion rate (%) = number of treatment courses completed/6 × 100

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No